CLINICAL TRIAL: NCT04249401
Title: Real-world Evidence for Non-valvular Atrial Fibrillation Patients Treated With Oral Anticoagulation in the Nordics
Brief Title: Study to Gather Information About the Safety of Oral Anticoagulation Drugs and How Well These Drugs Work in Real World for Patients With Non-valvular Atrial Fibrillation (Irregularly Heart Beats Which is Not Caused by a Heart Valve Problem)
Acronym: REATTAIN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: 20030
Record Dates: First submitted 2020-01-17; First posted 2020-01-31 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; apixaban; Dabigatran; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reduced dose NOAC: Participants with NVAF initiating treatment with reduced doses of individual non-vitamin K antagonist oral anticoagulants (NOACs)
  Interventions: Drug: Rivaroxaban (Xarelto); Drug: Apixaban; Drug: Dabigatran
- Vitamin K antagonists (VKA): Participants with NVAF initiating treatment with vitamin K antagonists (VKA)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto) — NOAC, reduced dose
  Groups: Reduced dose NOAC
Drug: Apixaban — NOAC, reduced dose
  Groups: Reduced dose NOAC
Drug: Dabigatran — NOAC, reduced dose
  Groups: Reduced dose NOAC
Drug: Warfarin — VKA
  Groups: Vitamin K antagonists (VKA)

SUMMARY:
Oral anticoagulant (OAC) treatment with either vitamin K antagonists (VKAs) or non-vitamin K antagonist oral anticoagulants (NOACs) is essential in patients with atrial fibrillation for the prevention of stroke or systemic embolism (SE) a condition that happens when a blood clot forms elsewhere in the body and travels through the blood stream to plug another vessel. While there are significant number of real-world publications on the use and outcomes of NOACs for stroke prevention, evidence from routine clinical practice on the use and outcomes of reduced doses of NOACs is scarce. By evaluating routine clinical practice data from national registers in Denmark, Finland, Norway and Sweden, researchers want to gather information about the safety and how well reduced doses of NOACs work in patients with irregularly heartbeats which are not caused by a heart valve problem (non-valvular atrial fibrillation, NVAF). As a primary aim of this study, treatment with low doses of NOACs (Xarelto [generic name rivaroxaban], Eliquis [generic name apixaban] or Pradaxa [generic name dabigatran]) will be compared with VKAs (warfarin) in Nordic patients with NVAF to assess the occurrence of stroke and systemic embolism [effectiveness]) and intracranial hemorrhage a type of bleeding that occurs inside the skull [safety]).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a qualifying oral OAC dispensed during the study period
* A primary diagnosis indicative of atrial fibrillation during the baseline period

Exclusion Criteria:

* Age < 18 years at index date
* Died on index date
* A diagnosis of valvular disease, pregnancy, transient cause of atrial fibrillation or venous thromboembolism in the baseline period or on the index date
* Hip or knee replacement surgery in the 60 days prior to or on the index date
* A dispensed prescription of heparin or fondaparinux in the 60 days prior to or on the index date
* A diagnosis of end-stage kidney disease or renal replacement therapy in the baseline period or on the index date
* More than one dispensed OAC (any dose of rivaroxaban, apixaban, dabigatran, edoxaban, or warfarin) on the index date
* A dispensed prescription of an OAC (any dose of rivaroxaban, apixaban, dabigatran, edoxaban, or warfarin) during the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NVAF who initiate treatment with oral anticoagulants (OACs, either VKAs or NOACs)
Sampling Method: Non-Probability Sample
Enrollment: 134897 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with ischemic stroke (IS) or systemic embolism (SE) | Retrospective analysis from 2010 - 2018
  Evaluation will be done in participants treated with reduced doses of individual NOACs and with VKA
Number of participants with intracranial haemorrhage (ICH) | Retrospective analysis from 2010 - 2018
  Evaluation will be done in participants treated with reduced doses of individual NOACs and with VKA

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.